CLINICAL TRIAL: NCT06070558
Title: ChAracterization of Normal and Pathological moRphological Variations of the TEMporomandibular Joint by Real-time magnetIc reSonance Imaging
Acronym: ARTEMIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Pedro TEIXEIRA-GONDIM, MD, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-A02648-33
Record Dates: First submitted 2023-07-10; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Healthy; Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy (Other): Healthy volunteers
  Interventions: Device: MRI with Real Time MRI Rapid Flash sequence
- Temporomandibular Joint Disorders (Other): Patients with Temporomandibular Joint Disorders
  Interventions: Device: MRI with Real Time MRI Rapid Flash sequence

INTERVENTIONS:
Device: MRI with Real Time MRI Rapid Flash sequence — MRI examination of temporomandibular joint with Real Time MRI Rapid Flash sequence

SUMMARY:
The Real Time MRI Rapid Flash sequence is particularly interesting for the study of moving organs and joints.

This sequence will make it possible to characterize normal and pathological temporomandibular joint movements by MRI.

ELIGIBILITY:
Inclusion Criteria:

* Adult: age ≥ 18 years old;
* Person with the capacity to understand the instructions given;
* Person affiliated to a social security scheme or beneficiary of such a scheme;
* Person having received complete information on the organization of the Clinical Investigation and having signed informed consent.

Exclusion Criteria:

* Person with large-scale metallic dental reconstructions;
* Edentulism more than 5 teeth;
* Claustrophobia;
* Contraindication to performing an MRI examination
* Persons referred to in Articles 64, 65 and 66 of European Regulation 2017/745 on Medical Devices (RDM) and in L. 1121-5 to L1121-8 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Curve representing the difference between displacement of condyles during Temporo Mandibular Joint (TMJ) movements in healthy subjects and in subjects with known Temporo Mandibular Disorder (TMD). | Baseline (day 0)

SECONDARY OUTCOMES:
Curve representing the displacement of the articular discs during TMJ movements | Baseline (day 0)
Curve representing the difference between displacement of joint discs during TMJ movements in healthy subjects and in subjects with known TMD | Baseline (day 0)
Characterization of the volume in mm3 of the main masticatory muscles during movement by MRI in healthy and pathological subjects. | Baseline (day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Nancy, Nancy, France